CLINICAL TRIAL: NCT02731157
Title: Rejuvesol® Washed RBC in Sickle Cell Patients Requiring Frequent Transfusions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: Pro00069955
Record Dates: First submitted 2016-04-02; First posted 2016-04-07 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2018-12

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Blood Transfusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Transfusion with rejuvenated red blood cells (RBCs) (Experimental): Subjects with sickle cell disease will receive RBCs treated with Rejuvesol®. Scheduled red cell exchanges performed with the last 4 units of the exchange having been incubated with Rejuvesol® solution. Only transfusions necessary for the treatment of the sickle cell disease will be given for the purpose of the study.
  Interventions: Drug: Rejuvesol; Procedure: Blood transfusion
- Transfusion with standard red blood cells (Active Comparator): Subjects with sickle cell disease will receive standard RBCs. Only transfusions necessary for the treatment of the sickle cell disease will be given for the purpose of the study.
  Interventions: Procedure: Blood transfusion

INTERVENTIONS:
Drug: Rejuvesol
  Arms: Transfusion with rejuvenated red blood cells (RBCs)
Procedure: Blood transfusion — Only transfusions necessary for the treatment of the sickle cell disease will be given for the purpose of the study.

SUMMARY:
The objective of this proposal is to test the feasibility of red blood cell (RBC) rejuvenation to chronic transfusion in sickle cell disease (SCD) and the potential benefit of RBC rejuvenation in this population to determine if a larger clinical trial powered to definitively characterize the benefits of rejuvenation is warranted.

This is a small pilot study is to see if restoring important energy molecules (ATP and 2,3,DPG) in stored red blood cells before they are transfused, with a rejuvenating solution (Rejuvesol), offers any advantages to individuals over standard blood transfusion. Subjects will receive either rejuvenated (R) or standard (S) RBCs with each transfusion for 6 transfusions (over approximately a 6-month period) in a pre-defined order to maximize detection of any signal.

DETAILED DESCRIPTION:
Blood transfusion is part of the standard care for individuals that have sickle cell disease. Often these transfusions become needed quite frequently. The purpose of the red blood cells in the blood is to deliver oxygen to the organs and tissues of the body. People with sickle cell disease have abnormal red blood cells. Stored blood undergoes some changes that may make it less effective in achieving this goal.

The purpose of this study is to see if restoring important energy molecules (ATP and 2,3,DPG) in stored red blood cells before they are transfused, with a rejuvenating solution (Rejuvesol), offers any advantages to individuals over standard blood transfusion. This is a Food and Drug Administration (FDA) approved process that is described by the American Association of Blood Banks for prolonging blood storage but not used for everyday transfusions. The investigators want to use this process to improve blood transfused to individuals who need frequent transfusions. Potential advantages include better delivery of oxygen by the transfused red blood cells and easier release of oxygen to the tissues. In addition the study will assess how using the rejuvenated blood affects the interval between transfusions. This means possibly that transfusions may not be needed as often.

Although Rejuvesol has been previously approved by the FDA, it is not routinely used to prepare standard blood transfusions to individuals who have sickle cell disease. Use of Rejuvesol in this study is considered investigational.

ELIGIBILITY:
Inclusion Criteria:

* Stable, compliant, chronically transfused sickle cell disease (SCD) patients
* Currently maintained crisis-free with repeated RBC therapy for at least 3 consecutive sessions
* ≥18 years old
* Have Hb SS disease
* Have the capacity to give informed consent

Exclusion Criteria:

* Baseline need for washed RBCs
* Pre-treatment SaO2 < 92%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian J Welsby, BSc MBBS, Principal Investigator — Duke University; Jay Raval, MD, Principal Investigator — University of North Carolina
Locations (2):
- United States (2):
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke Univeristy Medical Center, Durham, North Carolina

RESULTS

PARTICIPANT FLOW:
Groups:
- All Study Participants: Each participant in this 4 subject pilot study acted as their own control. Red cell exchanges (RCEs) occurred approximately every month and, over a 6 month period, the sequence of exchanges for each patient was: SRRRSS, where S=standard and R=rejuvenated RCEs.
Period: First Standard RCE
Arm/Group | All Study Participants
Started | 4
Completed | 4
Not Completed | 0
Period: First Rejuvenated RCE
Arm/Group | All Study Participants
Started | 4
Completed | 3
Not Completed | 1
Not completed — Withdrawal by Subject | 1
Period: Second Rejuvenated RCE
Arm/Group | All Study Participants
Started | 3
Completed | 3
Not Completed | 0
Period: Third Rejuvenated RCE
Arm/Group | All Study Participants
Started | 3
Completed | 3
Not Completed | 0
Period: Second Standard RCE
Arm/Group | All Study Participants
Started | 3
Completed | 3
Not Completed | 0
Period: Third Standard RCE
Arm/Group | All Study Participants
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Study Participants
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Average Percent Hemoglobin (HbA) Decrement Per Day
Description: The %HbA decrement is the current pre-treatment HbA - previous post treatment HbA in %. The average %HbA decrement per day was calculated using matched pairs.
Time Frame: 6 months
Population: Each participant acted as their own control with a sequence of rejuvenated and standard exchanges over 6 months. One subject ended further study participation after only 1 rejuvenated RBC exchange; limited data available.
Measure: Mean (Full Range); unit: %HbA per day
Groups:
- Transfusion With Rejuvenated Red Blood Cells (RBCs): Subjects with sickle cell disease will receive RBCs treated with Rejuvesol®. Scheduled red cell exchanges performed with the last 4 units of the exchange having been incubated with Rejuvesol® solution. Only transfusions necessary for the treatment of the sickle cell disease will be given for the purpose of the study.
  Rejuvesol
  Blood transfusion: Only transfusions necessary for the treatment of the sickle cell disease will be given for the purpose of the study.
Arm/Group | Transfusion With Rejuvenated Red Blood Cells (RBCs) | Transfusion With Standard Red Blood Cells
Number analyzed (Participants) | 4 | 4
%HbA per day | 0.629 [0.261 to 0.846] | 0.659 [0.261 to 0.846]
Statistical Analysis 1: Comparison: Transfusion With Rejuvenated Red Blood Cells (RBCs) vs Transfusion With Standard Red Blood Cells; Test type: Other; p = 0.95, ANOVA; Mean Difference (Final Values) = 0.65

2. Secondary Outcome: Actual HbA Decrement (g/dl) With Indexing to Calculated Circulating Blood Volume
Time Frame: 6 months
Population: Data not collected.
Arm/Group | Transfusion With Rejuvenated Red Blood Cells (RBCs) | Transfusion With Standard Red Blood Cells
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Actual HbA Decrement (g/dl) Without Indexing to Calculated Circulating Blood Volume
Time Frame: 6 months
Population: Data not collected.
Arm/Group | Transfusion With Rejuvenated Red Blood Cells (RBCs) | Transfusion With Standard Red Blood Cells
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in RBC Microparticles (MP) Counts
Time Frame: 6 months
Population: Data not collected.
Arm/Group | Transfusion With Rejuvenated Red Blood Cells (RBCs) | Transfusion With Standard Red Blood Cells
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in RBC/RBC-MP-mediated Thrombin Generation
Time Frame: 6 months
Population: Data not collected.
Arm/Group | Transfusion With Rejuvenated Red Blood Cells (RBCs) | Transfusion With Standard Red Blood Cells
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in p50 Pre- and Post-transfusion
Time Frame: 6 months
Population: Data not collected.
Arm/Group | Transfusion With Rejuvenated Red Blood Cells (RBCs) | Transfusion With Standard Red Blood Cells
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Transfusion With Standard RBCs: Each participant received three standard red cell exchanges.
- Transfusion With Rejuvenated RBCs: Each participant received three rejuvenated red cell exchanges.
Arm/Group | Transfusion With Standard RBCs | Transfusion With Rejuvenated RBCs
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-26): https://cdn.clinicaltrials.gov/large-docs/57/NCT02731157/Prot_SAP_000.pdf